CLINICAL TRIAL: NCT04426942
Title: Evaluation of the Couple's Sexuality During a Pregnancy Resulting From Medically Assisted Procreation and Comparison With Sexuality During a Spontaneous Pregnancy
Brief Title: Sexuality in Medically Assisted Procreation Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, Docteur, Central Hospital, Nancy, France
Other Study IDs: 2019PI2016
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Related; Assisted Reproduction
Keywords: assisted reproduction
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous pregnancy
  Interventions: Other: survey
- Assisted reproduction pregnancy
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — survey on sexuality during pregnancy

SUMMARY:
We wish to evaluate sexuality during pregnancy between spontaneous pregnancies and resulting from assisted procreation The literature is poor on thie subject

ELIGIBILITY:
Inclusion Criteria:

* physiological pregnancy
* pregnancy from assisted reproduction
* age over 18
* to understand french
* patient's agreement

Exclusion Criteria:

* pathological pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-06-20 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sexual functioning with Female Sexual Function Index (FSFI) test | In the second trimester of the pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Matthieu Dap, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided